CLINICAL TRIAL: NCT02369679
Title: Comparison of the Effectiveness of a Precast Adjustable Compression Wrap With the Multilayer Compression Bandage in Upper Limb Lymphedema
Brief Title: Effectiveness of Two Compression Methods in the Treatment of Upper Limb Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Germans Trias i Pujol Hospital (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Roser Belmonte, PhD, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/5584/I
Record Dates: First submitted 2015-02-04; First posted 2015-02-24 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Lymphedema
Keywords: upper limb; lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Precast Adjustable Compression Wrap (Experimental): Precast Adjustable Compression Wrap will be adjusted by the physiotherapist each visit
  Interventions: Device: Precast Adjustable Compression Wrap (Circaid)
- Multilayer Compression Bandages (Active Comparator): Multilayer Compression Bandages will be adjusted by the physiotherapist each visit
  Interventions: Device: Multilayer Compression Bandages

INTERVENTIONS:
Device: Precast Adjustable Compression Wrap (Circaid) — A physiotherapist well trained in lymphedema treatment will apply a lymphatic drainage to the affected upper limb. Then the physiotherapist will apply the precast adjustable compression wrap to the patient. The patient would maintain the precast adjustable compression wrap until the next session of treatment. The first 10 sessions will be daily from Monday to Friday.
  After the 10 first sessions, the treatment will be applied on alternate days (3 per week) until the patient receive a tailored compression garment (7-14 days).
  Arms: Precast Adjustable Compression Wrap
Device: Multilayer Compression Bandages — A physiotherapist well trained in lymphedema treatment will apply a lymphatic drainage to the affected upper limb. Then the physiotherapist will apply the multilayer bandage to the patient. The patient would maintain the multilayer compression bandage until the next session of treatment. The first 10 sessions will be daily from Monday to Friday.
  After the 10 first sessions, the treatment will be applied on alternate days (3 per week) until the patient receive a tailored compression garment (7-14 days).
  Arms: Multilayer Compression Bandages

SUMMARY:
Treatment of lymphedema is based on a combined program called complex decongestive therapy. The components of the complex decongestive therapy are skin care, kinesiotherapy, manual lymphatic drainage and compression. The compression with multilayer bandage has proved to be the most effective of these therapies when analyzed separately.The multilayer bandage produces a gradient compression on the limb where distal pressure is higher than proximal pressure. Several materials are needed for the multilayer bandage, including tubular bandage lining, digit bandages, foam under-cast padding and multiple layers of short-stretch bandages to cover the entire limb. The Precast Adjustable Compression Wrap fits each patient through a Velcro system.

The aim is to compare the effectiveness of a precast adjustable compression wrap (Circaid) with the multilayer compression bandages in the treatment of the upper limb lymphedema.

DETAILED DESCRIPTION:
The gold standard of the treatment of lymphedema is based on a combined program called complex decongestive therapy. The components of the complex decongestive therapy are skin care, kinesiotherapy, manual lymphatic drainage and compression. The compression with multilayer bandage has proved to be the most effective of these therapies when analyzed separately. With the multilayer compression bandage the upper limb lymphedema volume decreased a 37.2%.

The multilayer bandage produces a gradient compression on the limb where distal pressure is higher than proximal pressure. Several materials are needed for the multilayer bandage, including tubular bandage lining, digit bandages, foam under-cast padding and multiple layers of short-stretch bandages to cover the entire limb. The Precast Adjustable Compression Wrap fits each patient through a Velcro system.

Decreasing compression is achieved by controlling the tension applied to each Velcro through a visual color guide. The Precast Adjustable Compression Wrap has proved to be safe and effective to treat lower limb lymphedema, but there is little information about its effectiveness in the treatment of the upper limb lymphedema.

The aim is to compare the effectiveness of a precast adjustable compression wrap (Circaid) with the multilayer compression bandages in the treatment of the upper limb lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Upper limb lymphedema after axillary lymph node dissection for breast cancer.
* Lymphedema must affect at least the arm or the forearm.
* The lymphedema volume excess must be at least 10%
* The lymphedema must have not been previously treated or have been at least 1 year without treatment.

Exclusion Criteria:

* Bilateral upper limb lymphedema
* Cognitive or sensorial impairments which could interfere collaboration
* Plexopathy post radiotherapy
* Breast cancer in progression Pregnancy or Lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2016-01-19 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Change in the excess of volume of upper limb | Baseline to 3 months (10 sessions of treatment)
  Change in the excess of volume of the affected upper limb. The excess of volume is the difference in volume between the affected and the unaffected upper limb. The upper limb volumes will be obtained from the perimeters of the upper limbs and applying the truncate cone formula.
  Baseline to 2 weeks (10 sessions of treatment). A follow up at 3 months

SECONDARY OUTCOMES:
Changes in pain, heaviness, tightness and hardness | Baseline to 3 months (10 sessions of treatment)
  Changes in pain, heaviness, tightness and hardness will be measured by visual analogical scales. Baseline to 2 weeks (10 sessions of treatment). A follow up at 3 months
Changes in skin and lymphedema condition | Baseline to 3 months (10 sessions of treatment)
  The skin and lymphedema condition will be evaluated every day along the treatment phase and at 3 months of follow up. Baseline to 2 weeks (10 sessions of treatment). A follow up at 3 months
Number of Participants with Serious and Non-Serious Adverse Events | Baseline to 3 months (10 sessions of treatment)
  Collection of adverse effects spontaneously reported by the participants and/or observed by the investigators. In order to evaluate tolerability patients will be asked every day about any discomfort or troubles they could feel. On the other hand, it will be daily recorded how many hours the patient had used the precast adjustable compression wrap or the multilayer compression bandages. Baseline to 2 weeks (10 sessions of treatment). A follow up at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Roser Belmonte, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (3):
- Spain (3):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital Vall Hebron, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona